CLINICAL TRIAL: NCT03240354
Title: Reducing Intra-operative Pressure Variations in Paediatric Microcuff Endotracheal Tube Cuffs
Brief Title: Paediatric Microcuff Pressure Study
Acronym: MicroCuff
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nottingham University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17AN003
Record Dates: First submitted 2017-07-17; First posted 2017-08-07 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2018-03

CONDITIONS: Anesthesia; Pediatric; Intubation Complication

STUDY DESIGN:
Intervention Model Description: Prospective, blinded, randomised, parallel group control trial
Who Masked: Participant, Outcomes Assessor
Masking Description: * Participants will be split into two age groups, 'under 8 years' and '8 years and over', and a stratified randomisation method will be used to randomise each group, using a previously verified, sealed envelope, method and using blocks of unequal size.
  * Envelopes will be prepared using a random number table by an individual with no further role in the study
  * Each participant will be given a unique randomisation code matching the randomisation list
  * A record of each randomisation will be recorded on the Enrolment Log (TAFR01502)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Saline (Experimental): Use of saline to inflate cuff of endotracheal tube
  Interventions: Device: Saline cuff
- Control (Active Comparator): Use of air to inflate cuff of endotracheal tube
  Interventions: Device: Control

INTERVENTIONS:
Device: Saline cuff — Cuff of endotracheal tube inflated with saline rather than air (control)
  Arms: Saline
Device: Control — Cuff of endotracheal tube inflated with air
  Arms: Control

SUMMARY:
In paediatric anaesthesia, use of cuffed endotracheal (ET) tubes is subject to much debate. The concern is the possibility of damage to tracheal mucosa by excessive pressure from the cuff. The cuff pressure can increase during anaesthesia, especially if nitrous oxide is used.

Using saline to inflate the cuff has been shown to reduce intra-operative cuff pressure variation in adult studies, although it is not standard practice. Although the literature contains reports of cuff pressure increases during paediatric anaesthesia, there are no reports of attempts to address this. Use of pressure monitoring is recommended by AAGBI, but may not be consistently done. A safe method of limiting pressure, that is effective, imposes minimal extra workload and has minimal cost, would reduce risk to patients.

This study aims to investigate the effect on intra-operative cuff pressure of using saline to inflate the ET tube cuff, compared to standard practice of air inflation. Continuous pressure monitoring will be used to determine the proportion of cases where interventions are required to keep the pressure below a safe maximum level.

DETAILED DESCRIPTION:
During surgery under anaesthesia, use of cuffed endotracheal (ET) tubes is standard practice in adults. The cuff prevents air leak and protects the airway from soiling. Traditionally, in paediatric practice an uncuffed ET tube is used, sized according to the child's age. This prevents damage to the lining of the trachea by excessive pressure from the cuff.

The debate regarding the use of cuffed ET tubes in children is long-standing. New insight into the understanding of paediatric airway anatomy and newer designs of cuffed ET tubes (such as the MicroCuff Endotracheal tube, Halyard Health UK) have resulted in a shift towards their more frequent use. Studies suggest cuff pressures should be maintained below 20 - 25cm H2O, to minimise airway complications related to high pressures on the tracheal lining leading to inadequate blood flow, potentially causing swelling and, rarely, tracheal stenosis. This is of particular importance in small children, where even slight swelling can significantly reduce the airway diameter, with potentially serious consequences. Use of pressure monitoring is recommended by AAGBI, but may not be consistently done. A safe method of limiting pressure, that is effective, imposes minimal extra workload and has minimal cost, would reduce risk to patients.

The widespread use of nitrous oxide (N2O) in paediatric anaesthesia raises another issue. Nitrous oxide diffuses easily into the ET tube cuffs, raising the pressure within them. Various interventions have been trialled in adult studies to address this. Inflating ET tube cuffs with a mixture of air and N2O may be beneficial, but varying concentrations of N2O during anaesthesia limit the benefits. Filling the cuff with saline instead of air has been shown to prevent increases in cuff pressures in the adult population without any adverse safety issues, but it is still not standard practice.

Despite reports of similar variation in cuff pressures in paediatric patients, there have been no reported studies to date comparing the intra-operative changes in cuff pressures in children when the cuff is inflated with saline instead of air.

Therefore, the investigators propose to determine whether filling the ET tube cuff with saline prevents the changes in intra-cuff pressures, in children undergoing balanced anaesthesia with N2O, that are seen with air filled cuffs.

CLINICAL RELEVANCE The use of cuffed tubes in paediatric anaesthesia has become more and more common over the last decade. Newer, more anatomically based designs have helped to overcome many of the potential problems, but the issue of safe cuff pressures remains paramount.

Work in the adult literature has demonstrated the pressure at which there is a reduction in capillary perfusion. In paediatrics, the huge variation in capillary perfusion pressure makes finding an exact 'safe' level for every patient very difficult, but attempts have been made to characterise what an 'unsafe' level is.

The widespread use of nitrous oxide in paediatric anaesthesia also complicates the situation. The cuffs on modern paediatric cuffed tubes are very thin, allowing gasses to diffuse into them more easily. This means the volume (and thus the pressure) at the beginning of anaesthesia is not the same as at the end. Studies have also shown that the incidence of post-operative airway complications increases as the cuff pressure increases.

The AABGI has recently recommended cuff pressure monitoring as a minimum standard of care. However, achieving this through a lengthy case, where access to the airway may be limited, can prove challenging.

This studies hypothesis is that the use of saline, instead of air, in the cuff will lead to reduced pressure variation during anaesthesia, meaning that the pressure in the cuff at the end would be the same as at the beginning. This would minimise risk of complications for the patient and give a high level of patient safety and satisfaction, with minimal extra workload for the anaesthetist or expense for the NHS.

ELIGIBILITY:
Inclusion Criteria:

* Parent/guardian's written informed consent / age-appropriate participant assent
* Age: Birth to 16 years
* Elective surgery
* Endotracheal intubation with a cuffed tube required as part of general anaesthesia lasting longer than 45 minutes
* Planned use of N2O as part of balanced anaesthesia
* For questionnaire follow up; aged over 8 years without significant neurological impairment

Exclusion Criteria:

* Weight less than 3kg
* Laryngeal or tracheal pathology, including respiratory tract infections
* Difficulty in intubation (>2 attempts)
* NG tube placement during anaesthesia
* Nose, throat or airway surgery

Max Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 49 (Actual)
Dates: Start 2018-08-06 (Actual); Primary Completion 2019-07-30 (Actual); Study Completion 2019-07-30 (Actual)

PRIMARY OUTCOMES:
The number of cases where an intervention was required to maintain cuff pressure below 25cm H2O | Intra-operative, 45min - 6 hours
  * During anaesthesia, the pressure in the ET tube cuff will be measured continuously by an investigator, separate from the team providing the anaesthesia, using an arterial line pressure transducer set attached to the pilot balloon through a 3-way tap. The initial cuff pressure will be recorded ('Pressure 0')
  * The cuff pressure will be documented every 5 minutes.
  * If the cuff pressure exceeds 25 cm H2O for more than 30 seconds (to exclude artefactual changes), the volume of fluid in the cuff will be reduced until the pressure is returned to the initial level ('Pressure 0').
  * This constitutes an 'Intervention'

SECONDARY OUTCOMES:
Cuff pressure in each group | Intra-operative, 45min - 6 hours
  The mean cuff pressure for each patient will be calculated based on the recordings taken during the case
Post extubation adverse events | up to 20min Post extubation
  After removal of the ET tube at the end of the case, the attending anaesthetist will note any episodes of cough, stridor, laryngospasm, bradycardia of more than 10% from baseline or desaturation to below 92%, or by more than 10% from baseline. These will constitute a 'post extubation adverse event'
Post-operative airway complications | up to 24 hours post-op
  Post-operatively, prior to recovery discharge, children 8 years of age and over will be asked, by an observer blinded to their study group, to score any sore throat, dysphagia or hoarseness on a numerical rating scale.
  These questions will be asked again 8 - 24 hours post-operatively, prior to discharge home.

CONTACTS AND LOCATIONS:
Locations (1):
- Nottingham University Hospital, Nottingham, Nottinghamshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared outside the immediate research team

REFERENCES:
- [Background] Lonnqvist PA. Cuffed or uncuffed tracheal tubes during anaesthesia in infants and small children: time to put the eternal discussion to rest? Br J Anaesth. 2009 Dec;103(6):783-5. doi: 10.1093/bja/aep330. No abstract available. PMID 19918019
- [Background] Tobias JD. Pediatric airway anatomy may not be what we thought: implications for clinical practice and the use of cuffed endotracheal tubes. Paediatr Anaesth. 2015 Jan;25(1):9-19. doi: 10.1111/pan.12528. Epub 2014 Sep 20. PMID 25243638
- [Background] Weiss M, Dullenkopf A, Fischer JE, Keller C, Gerber AC; European Paediatric Endotracheal Intubation Study Group. Prospective randomized controlled multi-centre trial of cuffed or uncuffed endotracheal tubes in small children. Br J Anaesth. 2009 Dec;103(6):867-73. doi: 10.1093/bja/aep290. Epub 2009 Nov 3. PMID 19887533
- [Background] Suominen P, Taivainen T, Tuominen N, Voipio V, Wirtavuori K, Hiller A, Korpela R, Karjalainen T, Meretoja O. Optimally fitted tracheal tubes decrease the probability of postextubation adverse events in children undergoing general anesthesia. Paediatr Anaesth. 2006 Jun;16(6):641-7. doi: 10.1111/j.1460-9592.2005.01832.x. PMID 16719880
- [Background] Checketts MR, Jenkins B, Pandit JJ. Implications of the 2015 AAGBI recommendations for standards of monitoring during anaesthesia and recovery. Anaesthesia. 2017 Jan;72 Suppl 1:3-6. doi: 10.1111/anae.13736. No abstract available. PMID 28044335
- [Background] Dullenkopf A, Gerber AC, Weiss M. Nitrous oxide diffusion into tracheal tube cuffs: comparison of five different tracheal tube cuffs. Acta Anaesthesiol Scand. 2004 Oct;48(9):1180-4. doi: 10.1111/j.1399-6576.2004.00483.x. PMID 15352966
- [Background] Felten ML, Schmautz E, Delaporte-Cerceau S, Orliaguet GA, Carli PA. Endotracheal tube cuff pressure is unpredictable in children. Anesth Analg. 2003 Dec;97(6):1612-1616. doi: 10.1213/01.ANE.0000087882.04234.11. PMID 14633529
- [Background] Tu HN, Saidi N, Leiutaud T, Bensaid S, Menival V, Duvaldestin P. Nitrous oxide increases endotracheal cuff pressure and the incidence of tracheal lesions in anesthetized patients. Anesth Analg. 1999 Jul;89(1):187-90. doi: 10.1097/00000539-199907000-00033. PMID 10389801
- [Background] Karasawa F, Ohshima T, Takamatsu I, Ehata T, Fukuda I, Uchihashi Y, Satoh T. The effect on intracuff pressure of various nitrous oxide concentrations used for inflating an endotracheal tube cuff. Anesth Analg. 2000 Sep;91(3):708-13. doi: 10.1097/00000539-200009000-00040. PMID 10960405
- [Background] Combes X, Schauvliege F, Peyrouset O, Motamed C, Kirov K, Dhonneur G, Duvaldestin P. Intracuff pressure and tracheal morbidity: influence of filling with saline during nitrous oxide anesthesia. Anesthesiology. 2001 Nov;95(5):1120-4. doi: 10.1097/00000542-200111000-00015. PMID 11684980
- [Background] Bennett MH, Isert PR, Cumming RG. Postoperative sore throat and hoarseness following tracheal intubation using air or saline to inflate the cuff--a randomized controlled trial. Anaesth Intensive Care. 2000 Aug;28(4):408-13. doi: 10.1177/0310057X0002800409. PMID 10969368
- [Background] Tobias JD, Schwartz L, Rice J, Jatana K, Kang DR. Cuffed endotracheal tubes in infants and children: should we routinely measure the cuff pressure? Int J Pediatr Otorhinolaryngol. 2012 Jan;76(1):61-3. doi: 10.1016/j.ijporl.2011.09.033. Epub 2011 Oct 22. PMID 22024576
- [Background] Seegobin RD, van Hasselt GL. Endotracheal cuff pressure and tracheal mucosal blood flow: endoscopic study of effects of four large volume cuffs. Br Med J (Clin Res Ed). 1984 Mar 31;288(6422):965-8. doi: 10.1136/bmj.288.6422.965. PMID 6423162
- [Background] Sheraton TE, Gildersleve CD, Hall JE. The use of nitrous oxide in paediatric anaesthetic practice in the United Kingdom: a questionnaire survey. Anaesthesia. 2007 Jan;62(1):62-6. doi: 10.1111/j.1365-2044.2006.04857.x. PMID 17156228
- [Background] Constant I, Louvet N, Guye ML, Sabourdin N. [General anaesthesia in children: a French survey of practices]. Ann Fr Anesth Reanim. 2012 Sep;31(9):709-23. doi: 10.1016/j.annfar.2012.06.004. Epub 2012 Jul 7. French. PMID 22776772
- [Background] Calder A, Hegarty M, Erb TO, von Ungern-Sternberg BS. Predictors of postoperative sore throat in intubated children. Paediatr Anaesth. 2012 Mar;22(3):239-43. doi: 10.1111/j.1460-9592.2011.03727.x. Epub 2011 Nov 8. PMID 22066487
- [Derived] Armstrong J, Jenner P, Poulose S, Moppett IK. The effect of saline versus air for cuff inflation on the incidence of high intra-cuff pressure in paediatric MicroCuff(R) tracheal tubes: a randomised controlled trial. Anaesthesia. 2021 Nov;76(11):1504-1510. doi: 10.1111/anae.15493. Epub 2021 Apr 23. PMID 33891328